CLINICAL TRIAL: NCT00383357
Title: Aging, Hypnotics, Sleep Inertia and the Risk of Falling
Brief Title: Sleepiness and the Risk of Falling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AG0070; 5R03AG024621-02 (NIH); 5M01RR000051-45 (NIH)
Record Dates: First submitted 2006-09-28; First posted 2006-10-03 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Aging; Balance; Sleep
Keywords: Performance; Gait stability; sedative; hypnotic; quality of life; sleep disorder; wakefulness; sleeping pills; Cognitive function
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Zolpidem

INTERVENTIONS:
Drug: zolpidem

SUMMARY:
The purpose of this project is to examine the impact of sleeping pills and waking up in the middle of the night on walking balance and cognitive function, to identify risk factors for falls in older adults. A significant percentage of falls, approximately 33 to 52 percent, occur during the nighttime and morning hours when people are normally sleeping; therefore, it is possible that sleep and sleeping medication related impairments in balance may contribute to this risk.

DETAILED DESCRIPTION:
Awakening from sleep is well documented to impair cognitive performance in young adults. This phenomenon, called sleep inertia, has been reported to impair performance just as much as one night of total sleep deprivation, suggesting that there are significant functional consequences to sleep inertia. However, whether walking stability is impaired by sleep inertia is unknown. If sleep inertia impairs walking stability, it could be an important but currently unrecognized risk factor for falls in older adults. Also, the impact of aging on sleep inertia-related impairments in cognitive performance is unknown.

Sleeping medication use is higher in older than younger adults, and is a risk factor for falls. Current evidence suggests that sleeping medications impair walking stability and cognitive performance in young and older adults during wakefulness; however, no study has examined walking stability and cognitive performance of young and older adults upon awakening from sleep at night after taking a hypnotic (sleeping medication). Therefore, the purpose of this study is to determine whether sleep inertia and hypnotic use impairs walking stability and cognitive performance more in healthy older than in healthy younger adults. It is expected that findings from the proposed study will provide evidence for sleep inertia as a risk factor for falls in older adults.

Twelve older (aged 60-85) and twelve younger (aged 18-35) healthy male and female volunteers will participate in the study. The investigational procedures will include medical screening (e.g., physical, blood and urine tests, and bone mineral density assessment), home monitoring of sleep schedules for three weeks, and three overnight visits in the laboratory spaced approximately one week apart. During the laboratory visits, participants will be awakened in the middle of the night to perform walking stability and cognitive function tests. Before going to bed, participants will take either a placebo pill or a sleeping medication. On one of the visits, participants will be asked to go to bed about 2 hours later than usual.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Aged 18 to 35, or 60 to 85
* Lived at Denver altitude or higher for at least one year
* Stable treated diseases: thyroid dysfunction (including hypothyroidism and hyperthyroidism), hypertension, hypercholesterolemia, urinary incontinence, prostate enlargement, gastroesophageal reflux disease, irritable bowel syndrome

Exclusion Criteria:

* Aged 36 to 59, under 18, or over 85
* BMI less than 18.6 or greater than 30 kg/m2, women below 95 pounds regardless of BMI
* Sleep duration is less than 5 or more than 9 hours
* Sensitivity to sleeping medications
* Night work in the preceding 6 months
* Transmeridian travel (across more than 2 time zones) in the last 1 month
* Bone mineral density DXA T-score of less than -1.75
* Orthostatic intolerance
* Prior history of falls in past year
* Prior history of injurious fall in past 5 years
* Hip fracture following a fall
* Difficulty rising from a sitting position without use of hands to push off
* Needing to walk slowly or with a wide base of support to maintain balance
* Hormone replacement therapy for less than 3 months
* Connective Tissue and Joint Disorders
* Neurologic Disorders
* Musculoskeletal Disorders
* Immune Disorders
* Sleep Disorders
* Chronobiologic Disorders
* Cardiovascular Disorders
* Respiratory Disorders
* Kidney and Urinary Tract Disorders
* Infectious Diseases
* Gastrointestinal Disorders
* Hematopoietic Disorders
* Neoplastic Diseases
* Endocrine and Metabolic Diseases
* Psychopathology
* Dementia
* Drug dependency

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2004-08

PRIMARY OUTCOMES:
Changes in gait stability: normal walking and beam walking across force plates (platforms with sensors that measure the force (energy) that occurs when the foot contacts the ground during walking)
at 1, 15, and 30 minutes after awakening in the middle of the night during all three visits

SECONDARY OUTCOMES:
Changes in gait stability: normal walking and beam walking across force plates at 1, 15, and 30 minutes after awakening in the morning during all three visits.
cognitive performance: computerized assessment of executive function at 5, 20, and 35 minutes after awakening in the middle of the night and in the morning during all three visits.
sleep architecture: visual scoring of the sleep EEG across 8 hours of scheduled sleep during all three visits.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth P. Wright, PhD, Principal Investigator — Department of Integrative Physiology, University of Colorado; Danielle J. Frey, PT, MS, Study Director — Department of Integrative Physiology, University of Colorado
Locations (1):
- University of Colorado at Boulder, Boulder, Colorado, United States

REFERENCES:
- [Background] Brassington GS, King AC, Bliwise DL. Sleep problems as a risk factor for falls in a sample of community-dwelling adults aged 64-99 years. J Am Geriatr Soc. 2000 Oct;48(10):1234-40. doi: 10.1111/j.1532-5415.2000.tb02596.x. PMID 11037010
- [Background] Luukinen H, Koski K, Honkanen R, Kivela SL. Incidence of injury-causing falls among older adults by place of residence: a population-based study. J Am Geriatr Soc. 1995 Aug;43(8):871-6. doi: 10.1111/j.1532-5415.1995.tb05529.x. PMID 7636094
- [Background] Wertz AT, Ronda JM, Czeisler CA, Wright KP Jr. Effects of sleep inertia on cognition. JAMA. 2006 Jan 11;295(2):163-4. doi: 10.1001/jama.295.2.163. No abstract available. PMID 16403927
- [Derived] Frey DJ, Ortega JD, Wiseman C, Farley CT, Wright KP Jr. Influence of zolpidem and sleep inertia on balance and cognition during nighttime awakening: a randomized placebo-controlled trial. J Am Geriatr Soc. 2011 Jan;59(1):73-81. doi: 10.1111/j.1532-5415.2010.03229.x. PMID 21226678